CLINICAL TRIAL: NCT00314275
Title: Evaluation of Pharmacokinetics (PK) and Safety of the Medtronic Endeavor Drug (ABT-578) Eluting Coronary Stent System in De Novo Native Coronary Artery Lesions
Brief Title: The ENDEAVOR Pharmacokinetic (PK) Registry: The Medtronic Endeavor Drug Eluting Coronary Stent System
Acronym: ENDEAVOR PK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-061
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
Keywords: Pharmacokinetics; Coronary Artery Disease; PCI; Drug Eluting Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ENDEAVOR (Experimental): Drug Eluting Stent
  Interventions: Device: Coronary Artery Stenting; Device: Endeavor

INTERVENTIONS:
Device: Coronary Artery Stenting — Drug eluting stent
Device: Endeavor — Drug eluting stent

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) and safety associated with ABT-578 administered using the Medtronic Endeavor Drug Eluting Coronary Stent system in the treatment of single de novo lesions in native coronary arteries between 2.5 - 3.5 mm in diameter.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age.
* The patient has clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia, or a positive functional study.
* The patient is an acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting, and emergent coronary artery bypass graft (CABG) surgery.
* Female patients of childbearing potential must have a negative pregnancy test within 7 days before the procedure.
* The patient or patient's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board of the respective clinical site.

Exclusion Criteria:

* A known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, ticlopidine or clopidogrel, cobalt, nickel, chromium, molybdenum, polymer coatings, or a sensitivity to contrast media, which cannot be adequately pre-medicated.
* History of an allergic reaction or significant sensitivity to drugs similar to ABT-578, rapamycin, tacrolimus, everolimus, or any other analog or derivative.
* A platelet count < 100,000 cells/mm³ or > 700,000 cells/mm³, or a white blood cell (WBC) count < 3,000 cells/mm³.
* A creatinine level > 2.0 mg/dL within seven days prior to index procedure. Evidence of an acute myocardial infarction within 72 hours of the intended treatment (defined as: Q wave or non-Q wave myocardial infarction having creatine kinase [CK] enzymes greater than or equal to 2 X the upper laboratory normal with the presence of a creatine kinase myocardial-band isoenzyme [CK-MB] elevated above the institution's upper limit of normal).
* Previous percutaneous coronary intervention (PCI) of the target vessel within 9 months pre-procedure.
* Planned PCI of any vessel within 30 days post-procedure.
* During the index procedure, the target lesion requires treatment with a device other than PTCA prior to stent placement (such as, but not limited to: cutting balloon, directional coronary atherectomy, excimer laser, rotational atherectomy, thrombectomy, etc.).
* History of a stroke or transient ischemic attack within the prior 6 months. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months.
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Concurrent medical condition with a life expectancy of less than 12 months. Any previous or planned treatment of the target vessel with anti-restenotic therapies including, but not limited to, brachytherapy.
* Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints; or requires coronary angiography, intravascular ultrasound (IVUS) or other coronary artery imaging procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-01; Primary Completion 2006-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (Cmax, Tmax, AUC, T1/2, CL, etc.) | 9 months

SECONDARY OUTCOMES:
Success (device, lesion, and procedure) | 9 months
Major adverse cardiac event (MACE) rate | 30 days, 6, 9 and 12 months
Target site revascularization (TSR), target vessel revascularization (TVR), and target vessel failure (TVF) rate | 9 months
For patients receiving overlapping stents at the target lesion: angiographic parameters (in-stent and in-segment), including: late lumen loss | 8 months
Late loss index | 9 months
Angiographic binary restenosis (ABR) rate | 9 months
Minimum luminal diameter (MLD) | 9 months
Percent diameter stenosis (%DS) | 9 months
Neointimal hyperplastic volume as measured by intravascular ultrasound (IVUS) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, M.D., Principal Investigator — Columbia University
Locations (1):
- Santa Rosa Memorial Hospital, Santa Rosa, California, United States

REFERENCES:
- [Derived] Mauri L, Massaro JM, Jiang S, Meredith I, Wijns W, Fajadet J, Kandzari DE, Leon MB, Cutlip DE, Thompson KP. Long-term clinical outcomes with zotarolimus-eluting versus bare-metal coronary stents. JACC Cardiovasc Interv. 2010 Dec;3(12):1240-9. doi: 10.1016/j.jcin.2010.08.021. PMID 21232717